CLINICAL TRIAL: NCT00332514
Title: Post-Discharge Follow-Up Phone Call by a Pharmacist and Impact on Patient Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-23071
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2006-03

CONDITIONS: Readmission, Hospital
Keywords: pharmacist intervention; post-discharge telephone call; black hole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients offered follow-up phone call (Other): Patients offered follow-up telephone call
  Interventions: Behavioral: telephone call by a pharmacist

INTERVENTIONS:
Behavioral: telephone call by a pharmacist

SUMMARY:
The purpose is to analyze whether a follow-up telephone call by a pharmacist after patient discharge from the hospital can improve patient outcomes.

Patients will be interviewed via telephone within 72 hours of being discharged home from the hospital. Patients will be questioned on three main topics. They are:

1. Medical care
2. Medications
3. Follow-up appointments

The purpose is to find out if people understand discharge medications, have obtained those medications, are having any problems with their medications and have scheduled necessary follow-up appointments. It will be determined if a telephone call by a pharmacist will prevent patients from needing to go to the Emergency Room or being admitted back to the hospital.

DETAILED DESCRIPTION:
There is a time between hospital discharge and patient follow-up that has been deemed by many healthcare workers as a "black hole " (1). It is a time during which continuity of care is of utmost importance, yet there is no effective uniform system in place to ensure this vital continuity. During the post-discharge period (time from when the patient leaves the hospital to the time of first follow-up appointment), new medical problems can arise and old ones can be exacerbated. Additionally, patients can encounter innumerable barriers to healthcare, including difficulty obtaining medications and securing appointments with physicians or specialists. Also, patients may not have received proper counseling on new discharge medications, including proper use and potential side effects. Despite this important aspect of patient care, only a paucity of literature on the topic exists. Of the literature that does exist, it suggests that patient education concerning discharge planning and the post-discharge period is an aspect of care that is in great need of improvement and an excellent opportunity for intervention by a pharmacist.

This led to our research hypothesis, can a follow-up phone call from a pharmacist improve patient outcomes?

The primary endpoint of this study is a reduction in the number of hospital readmissions (any cause) during the 30-day post-discharge period. Thirty-day readmission rates will be compared to see if there is a difference between the intervention group (follow-up phone call) and control group (no phone call). The secondary outcomes include the number of patients in the study group for whom medication errors, complications or misuse could be identified.

References: (1). Kathuria, et al. Post-discharge follow-up: hospitalists dial into the "black hole". Hospitalist and Inpatient Management Report, June 2003

ELIGIBILITY:
Inclusion Criteria:

* admission to Internal Medicine Service on the Menino Pavilion, either Firm A or B at Boston Medical Center located in Boston, MA
* age greater than or equal to 18 years
* discharge to home from the inpatient General Medical Service
* English-speaking or lives with English-speaking person
* access to a working phone

Exclusion Criteria:

* admission to any other service at Boston Medical Center located in Boston, MA besides Internal Medicine Firms A or B
* age less than 18 years
* discharge to site other than home
* non-English-speaking or does not live with an English-speaking person
* no access to a working phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is a reduction in the number of hospital readmissions (any cause) during the 30-day post-discharge period.

SECONDARY OUTCOMES:
The secondary outcomes include the number of patients in the study group for whom medication errors, complications or misuse could be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Gail M Burniske, PharmD, BCPS, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States